CLINICAL TRIAL: NCT05561530
Title: A Phase 1/1b, Double-Blind, Randomized, Placebo-Controlled, First-in-Human Study of Subcutaneously Administered ALG-125755 to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Single Ascending Doses in Healthy Volunteers (Part 1) and Subjects With Chronic Hepatitis B (Part 2), and Multiple Doses in Subjects With Chronic Hepatitis B (Part 3)
Brief Title: A Study of ALG-125755 to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After Single Doses in Healthy Volunteers, and Single and Multiple Doses in CHB Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Single doses demonstrated an acceptable safety profile and antiviral activity at all doses evaluated.
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-125755-501
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALG-125755 (Experimental): Subcutaneous injections of ALG-125755 in HV or CHB subjects, up to 6 injections over the course of up to 72 weeks
  Interventions: Drug: ALG-125755
- Placebo (Placebo Comparator): Subcutaneous injections of placebo in HV or CHB subjects, up to 6 injections over the course of up to 72 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALG-125755 — single or multiple doses of ALG-125755
  Arms: ALG-125755
Drug: Placebo — single or multiple doses of placebo
  Arms: Placebo

SUMMARY:
A randomized study of ALG-125755 to evaluate safety, tolerability, pharmacokinetics, and pharmacodynamics after single doses in healthy volunteers, and single and multiple doses in CHB subjects

ELIGIBILITY:
Inclusion Criteria for All Subjects:

1. Female subjects must have a negative serum pregnancy test at screening
2. Subjects must have a 12-lead electrocardiogram (ECG) that meets the protocol criteria

Inclusion Criteria for Healthy Subjects:

1. Male or female between 18 and 55 years of age, extremes included.
2. Subjects must have a body mass index (BMI) of 18.0 to 32.0 kg/m2, extremes included.

Inclusion Criteria for CHB Subjects (Parts 2 and 3):

1. Subjects must be 18 to 70 years of age, inclusive of extremes.
2. Subjects may have a BMI of 18.0 to 35.0 kg/m2, extremes included.
3. For virally suppressed subjects, must be currently receiving HBV NA treatment for ≥6 months prior to screening. For currently not treated or treatment naïve subjects, must have never received treatment OR have not been on treatment within 6 months prior to randomization

Exclusion Criteria for All Subjects:

1. Subjects with any current or previous illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject or that could prevent, limit, or confound the protocol specified assessments or study results' interpretation
2. Subjects with a past history of cardiac arrhythmias, risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) or history or clinical evidence at screening of significant or unstable cardiac disease etc.
3. Subjects with a history of clinically significant drug allergy
4. Subject with current or history of clinically significant (as determined by the Investigator) skin disease requiring intermittent or chronic treatment
5. Excessive use of alcohol defined as regular consumption of

   ≥14 standard drinks/week for women and ≥21 standard drinks/week for men
6. Subjects with Hepatitis A, B, C, D, E or HIV-1/HIV-2 infection or acute infections such as SARS- CoV-2 infection

Exclusion Criteria for Healthy Volunteers (Part 1):

1. Unwilling to abstain from alcohol use for 48 hours prior to start of study through end of study follow up.
2. Subjects with renal dysfunction [e.g., estimated creatinine clearance <90 mL/min/1.73 m2 at screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula]

Exclusion criteria for CHB subjects (Parts 2 and 3):

1. Subjects who are positive for anti-HBs antibodies.
2. Subject with any history or current evidence of hepatic decompensation such as: variceal bleeding, spontaneous bacterial peritonitis, ascites, hepatic encephalopathy, or active jaundice (within the last year).
3. History or current evidence of cirrhosis.
4. Subjects with liver fibrosis that is classified as Metavir Score ≥F3 liver disease
5. Subjects must have absence of signs of hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events as assessed by DAIDS v2.1 of various doses of ALG-125755 in HV subjects and CHB subjects | Up to 32 days for Part 1
Incidence and severity of treatment emergent adverse events as assessed by DAIDS v2.1 | Up to 52 days for Part 2
Incidence and severity of treatment emergent adverse events as assessed by DAIDS v2.1 | Up to 616 days for Part 3

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose (0 hours) up to 616 days
  Pharmacokinetic parameters of ALG-125755 in plasma
Area under the concentration time curve [AUC] | Predose (0 hours) up to 616 days
  Pharmacokinetic parameters of ALG-125755 in plasma
Time to maximum plasma concentration [Tmax] | Predose (0 hours) up to 616 days
  Pharmacokinetic parameters of ALG-125755 in plasma
Antiviral activity of ALG-125755 as measured by quantitative changes in serum | Predose (0 hours) up to 616 days
  Pharmacokinetic parameters of ALG-125755 in plasma
Minimum plasma concentration (Cmin) | Predose (0 hours) up to 616 days
  Pharmacokinetic parameters of ALG-125755 in plasma
Change in HBsAg from baseline through up to 112 days from last dose in multiple dose HBV infected subjects | screening to up to 112 days

CONTACTS AND LOCATIONS:
Locations (4):
- MBAL Sveta Sofia EOOD, Dept of Internal Medicine with Gastroenterology Section, Sofia, Bulgaria
- PMSI Republican Clinical Hospital "t. Mosneaga", ARENSIA Exploratory Medicine Phase 1 Unit, Chisinau, Moldova
- New Zealand Clinical Research, Auckland, New Zealand
- National Institute for Infection Diseases, ARENSIA Exploratory Medicine S.R.L., Bucharest, Romania